CLINICAL TRIAL: NCT06264804
Title: Analysis of Factors Associated With Threatened Aspiration in Patients Undergoing Small-incision Lenticule Extraction (SMILE) : Prospective Study
Brief Title: Risk Factors for Progressive Suction Loss in Corneal Refractive Surgery
Status: Recruiting | Type: Observational
Sponsor: Yifeng Yu (Other)
Responsible Party: Sponsor-Investigator, Yifeng Yu, Deputy Chief Physician of Ophthalmology, Second Affiliated Hospital of Nanchang University
Organization: Second Affiliated Hospital of Nanchang University (Other)
Other Study IDs: [2023] No. 86
Record Dates: First submitted 2024-01-10; First posted 2024-02-20 (Actual); Last update posted 2024-04-02 (Actual); Status verified 2024-04

CONDITIONS: Refractive Surgery

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- progressive suction loss group: Progressive suction loss occurs during the SMILE procedure
- Normal group: There was no progressive suction during the SMILE procedure

SUMMARY:
The goal of this Prospective observational studiesis to Characteristics of progressive suction loss.

DETAILED DESCRIPTION:
The goal of this Prospective observational studiesis to Characteristics of progressive suction loss. The main question[s] it aims to answer are: • Characteristics of people who do not develop progressive aspiration Characteristics of people with progressive aspiration Participants will The differences between the two groups were compared

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years;
2. Stable refractive state in the last 2 years, with yearly change in refractive power ≤ 0.50 D;
3. Spherical power ≤ -10.00D, cylindrical power ≤ -3.00 D;
4. Best Corrected Visual Acuity (BCVA) ≥ 16/20;
5. No use of corneal contact lenses two weeks before surgery.

Exclusion Criteria:

1. Eye diseases or histories beyond myopia and astigmatism, such as keratoconus;
2. Previous eye surgeries or histories of systemic illnesses;
3. Severe mental disorders like generalized anxiety disorder, panic disorder, depression, psychosis, and bipolar disorder, impeding cooperation with the doctor.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: all
Sampling Method: Non-Probability Sample
Enrollment: 800 (Estimated)
Dates: Start 2024-02-16 (Actual); Primary Completion 2024-07-01 (Estimated); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
Identify risk factors for progressive suction loss | 2024-12-01
  Progressive suction loss, the precursors to the loss of suction are quite evident. This study involved reviewing surgical videos and classifying patients into normal and progressive suction loss groups based on diagnostic criteria for progressive suction loss proposed by Huang. The intruding gas, liquid, and conjunctival tissue were analyzed using the ImageJ image processing software. Progressive suction loss was classified into three groups based on severity: Group A, where bubbles and wet spots begin to appear at the contact area between the suction ring and the corneal edge; Group B, where the area of bubbles and wet spots increases, exceeding 5% of the contact area as analyzed by ImageJ, but not spreading to the corneal surface; Group C, where bubbles and wet spots spread to the corneal surface, even affecting the laser scanning area.

CONTACTS AND LOCATIONS:
Overall Officials: yifeng yu, Study Director — Second Affiliated Hospital of Nanchang University
Locations (1):
- Yuyifeng, Nanchang, Jiangxi, China

IPD SHARING:
Plan to Share IPD: Undecided